CLINICAL TRIAL: NCT04685434
Title: Validity and Reliability Study of "Shriners Hospital for Children Upper Extremity Evaluation" in Children With Rheumatic Disease
Brief Title: Validity and Reliability of "Shriners Hospital Upper Extremity Evaluation" in Children With Rheumatic Disease
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Physiotherapist, PhD Student, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC_34
Record Dates: First submitted 2020-12-12; First posted 2020-12-28 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Arm; Rheumatic Diseases; Child, Only
Keywords: rheumatic diseases; children; function
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients diagnosed with rheumatic diseases.: The Shriners Hospital for Children Upper Extremity Evaluation, the Jebsen-Taylor Hand Function Test, and the Childhood Health Assessment Questionnaire will be administered in children with rheumatic diseases. The Shriners Hospital for Children Upper Extremity Evaluation will be administered two weeks after the first examination and the results will be compared.
  Interventions: Other: Shriners Hospital for Children Upper Extremity Evaluation

INTERVENTIONS:
Other: Shriners Hospital for Children Upper Extremity Evaluation — The interventions are evaluating tools for the functional performance of the upper extremity.
  Other Names: Jebsen-Taylor Hand Function Test; Childhood Health Assessment Questionnaire

SUMMARY:
The most commonly used performance tests to evaluate upper extremity function in children diagnosed with rheumatic disease are the 9-hole peg test and Jebsen Taylor hand function tests. Although these tests have advantages such as being able to be applied in a short time, providing objective data, being easily applicable in the clinical environment, and being cost-effective, these tests are non-specific performance tests. Fine motor skills specific to rheumatic diseases, planned for children; There is no test battery that examines the mobility and position of each segment of the upper extremity during a function in detail.

The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based assessment approved for use in children with hemiplegic cerebral palsy. In addition to spontaneous functional movement, it also evaluates the dynamical position, grip, and release movements of the upper extremity segments. Approved with a total of 22 questions/tasks observed for children aged 3-18. While the evaluation takes about 15 minutes, it takes about 15-30 minutes for the participant to score after the evaluation. The test battery can be created with the materials found in the physiotherapy clinic and is therefore very practical in terms of cost. In addition, due to the video recording of the evaluation, it provides a detailed examination opportunity to the evaluator both during and after the evaluation. However, it is superior to other tests in terms of creating a patient archive due to video recording.

This study aimed to introduce SHUEE to the literature as a new assessment tool to be used in pediatric rheumatic pathologies.

It is planned to include 25 volunteer pediatric patients diagnosed with rheumatic diseases in the study. Intra-observer and inter-observer reliability of SHUEE in children with a rheumatic diagnosis will be evaluated. For validity, the Jebsen-Taylor Hand Function test and Childhood Health Assessment Questionnaire will be used.

DETAILED DESCRIPTION:
Various questionnaires and test batteries are available to evaluate the functional activities of the upper extremities in children with upper extremity involvement. Among these questionnaires and test batteries, there are different performance tests evaluating the grip, wrist, and elbow movements in the upper extremity due to rheumatic disease. In the literature, the most common performance tests used in children diagnosed with rheumatic disease are the 9-hole peg test and the Jebsen Taylor hand function tests. Although these tests have advantages such as being able to be applied in a short time, providing objective data, being easily applicable in the clinical environment, and being accessible in terms of cost, these tests are non-specific performance tests. There is no test battery that examines the mobility and position of each segment of the upper extremity during a function in detail for motor skills specific to children with rheumatic diseases.

The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based assessment validated for use in children with hemiplegic cerebral palsy. In addition to spontaneous functional movement, it also evaluates the dynamical position, grip, and release movements of the upper extremity segments. Approved with a total of 22 questions/tasks observed for children aged 3-18. While the evaluation takes about 15 minutes, it takes about 15-30 minutes for the participant to score after the evaluation. The test battery can be created with the materials found in the physiotherapy clinic and is therefore very practical in terms of cost.

SHUEE provides detailed information about the location of the upper extremity segments during the function. In addition, due to the video recording of the evaluation, it provides a detailed examination opportunity to the evaluator after the evaluation. However, it is superior to other tests in terms of creating a patient archive due to video recording.

This study aimed to introduce SHUEE to the literature as a new assessment tool to be used in pediatric rheumatic pathologies.

ELIGIBILITY:
Inclusion Criteria:

* To be in the 10-18 ages group (In order for the devices to comply with the minimum measurement criteria and to be able to cooperate with the study)
* Being diagnosed with rheumatic diseases at least 6 months ago with only upper extremity affected
* Unilateral upper extremity involvement

Exclusion Criteria:

* Having an acute pathology that could affect walking
* To be diagnosed with orthopedic/neurological pathology that will affect work and cooperation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the patients who applied to the pediatric rheumatology clinic in the university hospital
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Shriners Hospital Upper Extremity Evaluation | Baseline
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function. The outcome is the total score of the spontaneous functional analysis, dynamic positional analysis, and grasp/release analysis. Higher scores mean a better outcome.
Jebsen-Taylor Hand Function Test | Baseline
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL). The outcome is the sum of time taken for each sub-test, which is rounded to the nearest second. Lower scores mean a better outcome. Except for the subtest titled writing, all subtest scores should be under 10 seconds at least.
Shriners Hospital Upper Extremity Evaluation | after two weeks from baseline
  The Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) is a video-based tool for the assessment of upper extremity function. The outcome is the total score of the spontaneous functional analysis, dynamic positional analysis, and grasp/release analysis. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The Childhood Health Assessment Questionnaire | Baseline
  It is a self-report questionnaire and is said to measure both disability and discomfort in children with chronic arthritis. It assesses functional ability in 8 domains of physical function (30 items) for children between the ages of 6 months up to 18 years. Each item is scored on a four-point scale ranging from 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), 3 (unable to do). Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davids JR, Peace LC, Wagner LV, Gidewall MA, Blackhurst DW, Roberson WM. Validation of the Shriners Hospital for Children Upper Extremity Evaluation (SHUEE) for children with hemiplegic cerebral palsy. J Bone Joint Surg Am. 2006 Feb;88(2):326-33. doi: 10.2106/JBJS.E.00298. PMID 16452744
- [Background] Ozdogan H, Ruperto N, Kasapcopur O, Bakkaloglu A, Arisoy N, Ozen S, Ugurlu U, Unsal E, Melikoglu M; Paediatric Rheumatology International Trials Organisation. The Turkish version of the Childhood Health Assessment Questionnaire (CHAQ) and the Child Health Questionnaire (CHQ). Clin Exp Rheumatol. 2001 Jul-Aug;19(4 Suppl 23):S158-62. PMID 11510322
- [Background] Sigirtmac IC, Oksuz C. Investigation of reliability, validity, and cutoff value of the Jebsen-Taylor Hand Function Test. J Hand Ther. 2021 Jul-Sep;34(3):396-403. doi: 10.1016/j.jht.2020.01.004. Epub 2020 Mar 7. PMID 32156578